CLINICAL TRIAL: NCT02301143
Title: Nab-paclitaxel (Abraxane) Plus Gemcitabine in Subjects With Locally Advanced Pancreatic Cancer (LAPC): An International, Open-label, Multi-center, Phase 2 Study (LAPACT).
Brief Title: Phase 2 Nab® -Paclitaxel (Abraxane®) Plus Gemcitabine in Subjects With Locally Advanced Pancreatic Cancer (LAPC)
Acronym: LAPACT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABI-007-PANC-007
Record Dates: First submitted 2014-11-14; First posted 2014-11-25 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Pancreatic Neoplasms
Keywords: Pancreatic Neoplasms; Pancreatic Cancer; Locally advanced pacriatic cancer; nab-Paclitaxel; Abraxane; Gemcitabine; ABI-007
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine; Chemoradiotherapy; Capecitabine; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- nab-Paclitaxel plus Gemcitabine (Experimental): nab-Paclitaxel 125 mg/m2 intravenous (IV) infusion over approximately 30 to 45 minutes on Days 1, 8, and 15, followed by gemcitabine 1000 mg/m2 IV infusion over approximately 30 minutes on Days 1, 8, and 15 of each 28-day cycle Subjects who complete 6 cycles of nab-paclitaxel and gemcitabine without disease progression or unacceptable toxicities, the Investigator will then determine the best option for the subject.
  * Continuation of nab-paclitaxel and gemcitabine therapy to disease progression or unacceptable toxicity OR
  * Chemoradiation therapy consisting of the concurrent use of capecitabine or gemcitabine with radiation according to institutional practice OR
  * Surgical intervention
  Interventions: Drug: nab-Paclitaxel; Drug: Gemcitabine; Drug: Chemoradiation; Drug: Capecitabine; Procedure: Surgery

INTERVENTIONS:
Drug: nab-Paclitaxel
  Other Names: Abraxane
Drug: Gemcitabine
  Other Names: Gemzar
Drug: Chemoradiation
Drug: Capecitabine
Procedure: Surgery — Surgical intervention

SUMMARY:
This clinical study is in subjects who are 18 years old or older with locally advanced pancreatic cancer who have not received prior treatment for their pancreatic cancer. The study treats all subjects with nab-Paclitaxel plus gemcitabine for approximately 6 months of treatment. Subjects who complete the treatment will choose, with their treating physicians, what additional treatment should be given: more nab-Paclitaxel plus gemcitabine, Chemoradiation therapy, or surgery to treat the locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
This is an international, non-randomized, open-label, multi-center, Phase 2 study in subjects who are 18 years old or older with locally advanced pancreatic cancer who have not received prior treatment for their pancreatic cancer. All subjects will be treated with nab-paclitaxel plus gemcitabine for 6 cycles followed by an Investigator's Choice of continuation of treatment with nab-paclitaxel plus gemcitabine, chemoradiation therapy, or surgery.

Safety assessments by laboratory testing and physical exams will be conducted through-out the study.

Efficacy assessments by physical exam will be preformed through-out the study and tumor imaging will be conducted approximately every 2 months.

Subjects will be considered active study participants from enrollment up to, but not including, survival follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Non- metastasis, unresectable, adenocarcinoma pancreatic cancer patients
* No prior anticancer therapy for pancreatic cancer

  •≥ 18 years of age with a performance status of 0 or 1•Adequate complete blood counts, hepatic function, and renal function
* Signed informed Consent

Exclusion Criteria:

* Active bacterial, viral, or fungal infection
* Infection with hepatitis B or C, or history of human immunodeficiency virus (HIV) infection, or receiving immunosuppressive or myelosuppressive
* Subjects with sensory neuropathy, ascites, or plastic biliary stent.
* Serious medical risk factors involving any of the major organ systems, or serious psychiatric disorders (including but not limited to connective tissue disorders, lung disease, and cardiac or seizure disorders)
* Women who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2015-04-21 (Actual); Primary Completion 2017-11-21 (Actual); Study Completion 2018-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teng Jin Ong, MD, Study Director — Celgene
Locations (42):
- United States (23):
  - Mayo Clinic - Arizona, Scottsdale, Arizona
  - UC Davis Cancer Center, Sacramento, California
  - Scripps Clinic Torrey Pines, San Diego, California
  - Smilow Cancer Hospital At Yale-New Haven, New Haven, Connecticut
  - Georgetown University Medical Center Lombardi Cancer Center, Washington D.C., District of Columbia
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Piedmont Cancer Institute PC, Atlanta, Georgia
  - Cancer Treatment Centers of America - Southeastern Regional Medical Center, Newnan, Georgia
  - ME Center for Cancer Medicine, Scarborough, Maine
  - Tufts - New England Medical Center, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - Saint Joseph Mercy Ann Arbor Hospital, Ann Arbor, Michigan
  - Karmanos Cancer Center Wayne State University, Detroit, Michigan
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Regional Cancer Care Associates LLC, Morristown, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Clinical Research Alliance, Lake Success, New York
  - State University of New York Upstate Medical Center, Syracuse, New York
  - Montefiore Einstein Cancer Center, The Bronx, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Mark H Zangmeister Center, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Houston Methodist Cancer Center, Houston, Texas
- Canada (5):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - CHUM Hôpital Saint-Luc, Montreal, Quebec
  - McGill University, Montreal, Quebec
- France (6):
  - Centre Regional de lutte contre le cancer Paul Papin, Angers
  - CHRU Besancon, Besançon
  - Centre Hospitalier Belfort Montbeliard, Besançon
  - Hopital Beaujon, Clichy
  - Hopital Saint Antoine, Paris
  - Hopital Haut Leveque, Pessac
- Italy (3):
  - Ospedale Sacro Cuore di Gesu FatebeneFratelli, Benevento
  - Azienda Ospedaliera Universitaria San Martino, Genova
  - Policlinico Universitario Campus Biomedico Di Roma, Roma
- Spain (5):
  - Hospital Universitario a Coruna, A Coruña
  - ICO-Hospital Germans Trias i Pujol, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Miguel Servet, Zaragoza

REFERENCES:
- [Derived] Philip PA, Lacy J, Portales F, Sobrero A, Pazo-Cid R, Manzano Mozo JL, Kim EJ, Dowden S, Zakari A, Borg C, Terrebonne E, Rivera F, Sastre J, Bathini V, Lopez-Trabada D, Asselah J, Saif MW, Shiansong Li J, Ong TJ, Nydam T, Hammel P. Nab-paclitaxel plus gemcitabine in patients with locally advanced pancreatic cancer (LAPACT): a multicentre, open-label phase 2 study. Lancet Gastroenterol Hepatol. 2020 Mar;5(3):285-294. doi: 10.1016/S2468-1253(19)30327-9. Epub 2020 Jan 14. PMID 31953079

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 152 patients were screened and 107 participants enrolled.
Groups:
- Nab-Paclitaxel Plus Gemcitabine: nab-Paclitaxel 125 mg/m^2 intravenous (IV) infusion administered over approximately 30-45 minutes on Days 1, 8, and 15, followed by gemcitabine 1000 mg/m^2 IV infusion over approximately 30 minutes on Days 1, 8, and 15 of each 28-day cycle for 6 cycles. For participants who completed 6 cycles of nab-paclitaxel and gemcitabine without disease progression or unacceptable toxicities, the Investigator then determined the best option for the participant in the Investigator's Choice Period.
- Investigator Choice: For participants who completed 6 cycles of nab-paclitaxel and gemcitabine without disease progression or unacceptable toxicities, the Investigator then determined the best option for the participant in the Investigator's Choice Period. Investigator Choice includes 3 options: 1. Continued on nab-Paclitaxel and gemcitabine 2. Chemoradiation 3. Surgical Intervention
Period: Induction Period
Arm/Group | Nab-Paclitaxel Plus Gemcitabine | Investigator Choice
Started (Participants enrolled.) | 107 | 0
Completed | 62 | 0
Not Completed | 45 | 0
Not completed — Enrolled But Not Treated | 1 | 0
Not completed — Death | 1 | 0
Not completed — Adverse Event | 22 | 0
Not completed — Progressive Disease | 8 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Noncompliance with Study Drug | 1 | 0
Not completed — Physician Decision | 4 | 0
Not completed — Symptomatic Deterioration | 2 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Other | 1 | 0
Period: Investigator's Choice
Arm/Group | Nab-Paclitaxel Plus Gemcitabine | Investigator Choice
Started | 0 | 47 (12 participants continued nab-Paclitaxel/Gemcitabine; 18 started chemoradiation;17 underwent surgery)
Completed | 0 | 37 (3 participants completed nab-Paclitaxel+Gemcitabine,18 completed chemoradiation,16 had surgery.)
Not Completed | 0 | 10
Not completed — Adverse Event | 0 | 3
Not completed — Progressive Disease | 0 | 3
Not completed — Noncompliance With Study Drug | 0 | 1
Not completed — Symptomatic Deterioration | 0 | 1
Not completed — Other | 0 | 1
Not completed — Unresectable Surgery | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population at start of Induction
Groups:
- Nab-Paclitaxel Plus Gemcitabine: In the Induction period, nab-paclitaxel 125 mg/m^2 intravenous (IV) infusion was administered over approximately 30-45 minutes on Days 1, 8, and 15, followed by gemcitabine 1000 mg/m^2 IV infusion over approximately 30 minutes on Days 1, 8, and 15 of each 28-day cycle. For participants who completed 6 cycles of nab-paclitaxel and gemcitabine without disease progression or unacceptable toxicities, the Investigator then determined the best option for the participant in the Investigator's Choice Period: - Continuation of nab-paclitaxel and gemcitabine therapy to disease progression or unacceptable toxicity OR - Chemoradiation therapy consisting of the concurrent use of capecitabine or gemcitabine with radiation according to institutional practice OR - Surgical intervention
Arm/Group | Nab-Paclitaxel Plus Gemcitabine
Number analyzed (Participants) | 107
Age, Continuous [Median (Full Range); unit: years] | 65.0 [42 to 85]
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 44
  >=65 - 75 years | 50
  >75 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 78
  Unknown or Not Reported | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 72
  More than one race | 0
  Unknown or Not Reported | 30
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status assesses how the disease affects the daily living activities of the participant and helps determine appropriate treatment and prognosis. - 0 = Fully Active (Most Favorable Activity); - 1 = Restricted activity but ambulatory; - 2 = Ambulatory but unable to carry out work activities; - 3 = Limited Self-Care; - 4 = Completely Disabled.
  Participants
    Grade 0 | 50
    Grade 1 | 57
    Grade 2 | 0
    Grade 3 | 0
    Grade 4 | 0
Physician Assessment of Peripheral Neuropathy [Count of Participants; unit: Participants] — Physician assessment for grading of peripheral neuropathy in participants receiving chemotherapy according to National Cancer Institute Common Toxicity Criteria (NCICTC): Grade 0 = None or no neuromotor or neurosensory loss; Grade 1 = Asymptomatic: loss of deep tendon reflexes or paresthesia; - Grade 2 = Moderate symptoms: limiting instrumental Activities of Daily Living (ADLs); - Grade 3 = Severe symptoms: limiting self-care ADL; assistance device indicated; - Grade 4 = Life-threatening consequences: urgent intervention indicated.
  Participants
    Grade 0 | 101
    Grade 1 | 6
    Grade 2 | 0
    Grade 3 | 0
    Grade 4 | 0
Baseline Albumin [Median (Full Range); unit: g/L] | 39.0 [28 to 50]
Carbohydrate Antigen 19-9 (CA19-9) [Median (Full Range); unit: U/mL] — Serum CA 19-9 concentrations may be elevated in patients with gastrointestinal malignancies such as pancreatic cancer. Population: Baseline CA19-9 measures are missing for six participants.
  U/mL
    number analyzed (Participants) | 101
    (all) | 243.3 [0 to 20741]
Baseline Neutrophil - to - Lymphocyte Ratio (NLR) [Count of Participants; unit: Participants] — Neutrophil to lymphocyte ratio (NLR) is used as a marker of subclinical inflammation. Increased NLR is associated with poor prognosis in advanced pancreatic cancer.
  Participants
    <= 5 | 91
    > 5 | 14
    Missing | 2
Sum of Longest Diameter of Target Lesions [Median (Full Range); unit: mm] | 44.0 [17 to 130]
Number of Target Lesions [Median (Full Range); unit: lesions] | 1.0 [1 to 3]
Time from Primary Diagnosis to First Dose [Median (Full Range); unit: days] | 27.0 [4 to 95]

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Estimates for Time to Treatment Failure (TTF)
Description: TTF was defined as the time after the first dose of study therapy to discontinuation of study therapy due to disease progression, death by any cause, or the start of a new non-protocol-defined anticancer therapy/surgery. If a participant does not progress, die or start a new non-protocol-defined anticancer therapy, the participant was censored on the last tumor assessment date.
  Tumor evaluations of CT or MRI scans were assessed by the investigative sites and response determined according to Response Evaluation Criteria in Solid Tumors (RECIST) guidelines, version 1.1.
  The definition for progressive disease (PD) was >= 20% increase in the sum of diameters of target lesions from nadir, and the sum showed an absolute increase of >= 5 mm; the progression of a non-target lesion or the appearance of any new lesions is also considered progression.
  Median and its 90% confidence interval (CI) of TTF were estimated using the method of Brookmeyer and Crowley.
Time Frame: Day 1 of study treatment up to 28.75 months; (maximum time for the last tumor assessment)
Population: Intent to treat population was defined as all participants enrolled into the study.
Measure: Median (90% Confidence Interval); unit: months
Groups:
- Nab-Paclitaxel Plus Gemcitabine: nab-Paclitaxel 125 mg/m^2 intravenous (IV) infusion administered over approximately 30-45 minutes on Days 1, 8, and 15, followed by gemcitabine 1000 mg/m^2 IV infusion over approximately 30 minutes on Days 1, 8, and 15 of each 28-day cycle. For participants who completed 6 cycles of nab-paclitaxel and gemcitabine without disease progression or unacceptable toxicities, the Investigator then determined the best option for the participant in the Investigator's Choice Period. - Continuation of nab-paclitaxel and gemcitabine therapy to disease progression or unacceptable toxicity OR - Chemoradiation therapy consisting of the concurrent use of capecitabine or gemcitabine with radiation according to institutional practice OR - Surgical intervention
Arm/Group | Nab-Paclitaxel Plus Gemcitabine
Number analyzed (Participants) | 107
months | 9.0 [7.26 to 10.05]

2. Secondary Outcome: Disease Control Rate (DCR): Percentage of Participants With Complete (CR) or Partial Response (PR), or Stable Disease (SD) for ≥ 16 Weeks According to RECIST Version 1.1
Description: DCR was defined as the percentage of participants with a CR or PR or SD from of date of first treatment to 16 weeks. Tumor assessments after start of non-protocol-defined anticancer therapy were excluded.
  RECIST 1.1 Definition:
  * CR: disappearance of all target and non-target lesions; any pathological lymph nodes (target or non-target) must have reduction in short axis to < 10 mm and no new lesions diagnosed.
  * PR: a >= 30% decrease in the sum of diameters of target lesions from baseline; no evidence of progression in any of the non-target lesions diagnosed at baseline; and no new lesions diagnosed.
  * SD: neither sufficient shrinkage to qualify for PR nor sufficient increase of lesions to qualify for PD.
  The two-sided 90% binomial confidence intervals (CIs) were estimated by Wilson score method.
Time Frame: Day 1 of study treatment up to the end of investigator choice period plus 28 days; up to 76.9 weeks
Population: Intent to treat population was defined as all participants enrolled into the study.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Nab-Paclitaxel Plus Gemcitabine
Number analyzed (Participants) | 107
percentage of participants | 77.6 [70.3 to 83.5]

3. Secondary Outcome: Overall Response Rate (ORR): Percentage of Participants With Complete (CR) or Partial Response (PR) According to RECIST Version 1.1
Description: ORR was defined as the percentage of participants that achieved a combined incidence of complete (CR) and partial response (PR) using RECIST 1.1 guidelines as assessed by the investigator. Assessments after new non-protocol-defined anticancer therapy are excluded. For participants who had resectable surgery in Investigator Choice period, assessments after surgical intervention are excluded.
  RECIST 1.1 Definition:
  * CR: disappearance of all target and non-target lesions; any pathological lymph nodes (target or non-target) must have reduction in short axis to < 10 mm and no new lesions diagnosed.
  * PR: a >= 30% decrease in the sum of diameters of target lesions from baseline; no evidence of progression in any of the non-target lesions diagnosed at baseline; and no new lesions diagnosed.
  The two-sided 90% binomial confidence intervals (CIs) were estimated by Wilson score method
Time Frame: Day 1 of study treatment up to the end of investigator choice period plus 28 days; up to 76.9 weeks
Population: Intent to treat population was defined as all participants who were enrolled into the study.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Nab-Paclitaxel Plus Gemcitabine
Number analyzed (Participants) | 107
percentage of participants | 39.3 [31.8 to 47.2]

4. Secondary Outcome: Kaplan-Meier Estimate of Progression-Free Survival (PFS)
Description: Progression-free Survival (PFS) was defined as the time from the date of the first dose to the date of disease progression or death (by any cause), whichever is earlier. The analysis day was calculated from enrollment date for one participant who was not treated. Participants who have no disease progression or have not died were censored to last tumor assessment date with progression-free.
  The definition for progressive disease (PD) was at least a 20% increase in the sum of diameters of target lesions from nadir; the sum must also demonstrate an absolute increase of >= 5 mm; the progression of a non-target lesion or the appearance of any new lesions is also considered progression.
  Median and its 90% confidence interval of PFS were estimated using the method of Brookmeyer and Crowley.
Time Frame: Day 1 of study treatment up to 28.75 months (maximum time for the last tumor assessment)
Population: Intent to treat population was defined as all participants who were enrolled into the study.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Nab-Paclitaxel Plus Gemcitabine
Number analyzed (Participants) | 107
months | 10.9 [9.26 to 11.63]

5. Secondary Outcome: Kaplan-Meier Estimates for Overall Survival (OS)
Description: Overall survival was defined as the time from the date of first dose of study therapy to the date of death (by any cause). Participants who were alive at the end of study or clinical data cut were censored on the last known time that the participant was alive or the clinical cutoff date, whichever was earlier. Median and its 90% confidence interval of OS were estimated using the method of Brookmeyer and Crowley
Time Frame: Day 1 of study treatment up to 31.34 months (maximum time for survival follow-up)
Population: Intent to treat population was defined as all participants who were enrolled into the study.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Nab-Paclitaxel Plus Gemcitabine
Number analyzed (Participants) | 107
months | 18.8 [14.95 to 24.02]

6. Secondary Outcome: Participant Counts in Response Categories Using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30): Global Health Status and 5 Functioning Scales
Description: The European Organization for Research and Treatment of Cancer Quality-of-Life questionnaire (EORTC QLQ-C30) is a validated health-related quality of life (HRQoL) measure. The EORTC QLQ-C30 is composed of both multi-item scales and single-item measures, including 5 functional scales, 3 symptom scales, 6 single symptom items, and 1 global health status / quality of life scale. No item occurs in more than one scale. All reported measures are transformed to a 0 - 100 scale. In the Global Health Status and 5 functional scales, 0 = worst possible quality of life/health status and 100 = best possible quality of life/health status. The best score on treatment is the best score from all post-baseline visits and is compared to the baseline to get the following responder categories. Responder categories: - Improved: >=10 increase from baseline - Stable: neither increase nor decrease >10 - Worsened: >=10 decrease from baseline
Time Frame: Baseline (Day -1), Day 1 of each cycle, for up to 19 cycles each cycle consisting of 28 days and the 28-day follow-up visit
Population: Intent to treat population was defined as all participants enrolled into the study with both baseline and post baseline values.
Measure: Count of Participants; unit: Participants
Groups:
- Nab-Paclitaxel Plus Gemcitabine: nab-Paclitaxel 125 mg/m^2 intravenous (IV) infusion administered over approximately 30-45 minutes on Days 1, 8, and 15, followed by gemcitabine 1000 mg/m^2 IV infusion over approximately 30 minutes on Days 1, 8, and 15 of each 28-day cycle. For participants who completed 6 cycles of nab-paclitaxel and gemcitabine the Investigator then determined the best option for the participant in the Investigator's Choice Period. - Continuation of nab-paclitaxel and gemcitabine therapy to disease progression or unacceptable toxicity OR - Chemoradiation therapy consisting of the concurrent use of capecitabine or gemcitabine with radiation according to institutional practice OR - Surgical intervention - Continuation of nab-paclitaxel and gemcitabine therapy to disease progression or unacceptable toxicity OR - Chemoradiation therapy consisting of the concurrent use of capecitabine or gemcitabine with radiation according to institutional practice OR - Surgical intervention
Arm/Group | Nab-Paclitaxel Plus Gemcitabine
Number analyzed (Participants) | 95
Participants
  Global Health Status: Improved | 43
  Global Health Status: Stable | 34
  Global Health Status: Worsened | 18
  Physical Functioning Scale: Improved | 20
  Physical Functioning Scale: Stable | 66
  Physical Functioning Scale: Worsened | 9
  Role Functioning Scale: Improved | 36
  Role Functioning Scale: Stable | 46
  Role Functioning Scale: Worsened | 13
  Emotional Functioning Scale: Improved | 50
  Emotional Functioning Scale: Stable | 40
  Emotional Functioning Scale: Worsened | 5
  Cognitive Functioning Scale: Improved | 33
  Cognitive Functioning Scale: Stable | 51
  Cognitive Functioning Scale: Worsened | 11
  Social Functioning Scale: Improved | 38
  Social Functioning Scale: Stable | 43
  Social Functioning Scale: Worsened | 14

7. Secondary Outcome: Participant Counts in Response Categories Using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30): Symptom Scales and Single Symptom Items
Description: The European Organization for Research and Treatment of Cancer Quality-of-Life questionnaire (EORTC QLQ-C30) is a validated health-related quality of life (HRQoL) measure. The EORTC QLQ-C30 is composed of both multi-item scales and single-item measures, including 5 functional scales, 3 symptom scales, 6 single symptom items, and 1 global health status / quality of life scale. No item occurs in more than one scale. All reported measures are transformed to a 0 to 100 scale. In the symptom scales and single symptom items, 0 = optimal health state and 100 = worst possible health state. The best score on treatment is the best score from all post-baseline visits and is compared to the baseline to get the following responder categories. Responder categories: - Improved: >=10 decrease from baseline - Stable: neither increase nor decrease >10 - Worsened: >=10 increase from baseline
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Groups:
- Nab-Paclitaxel Plus Gemcitabine: nab-Paclitaxel 125 mg/m^2 intravenous (IV) infusion administered over approximately 30-45 minutes on Days 1, 8, and 15, followed by gemcitabine 1000 mg/m^2 IV infusion over approximately 30 minutes on Days 1, 8, and 15 of each 28-day cycle. For participants who completed 6 cycles of nab-paclitaxel and gemcitabine, the Investigator then determined the best option for the participant in the Investigator's Choice Period. - Continuation of nab-paclitaxel and gemcitabine therapy to disease progression or unacceptable toxicity OR - Chemoradiation therapy consisting of the concurrent use of capecitabine or gemcitabine with radiation according to institutional practice OR - Surgical intervention
Arm/Group | Nab-Paclitaxel Plus Gemcitabine
Number analyzed (Participants) | 95
Participants
  Symptom Scale-Fatigue: Improved | 46
  Symptom Scale-Fatigue: Stable | 24
  Symptom Scale-Fatigue: Worsened | 25
  Scale-Nausea+Vomiting: Improved | 29
  Scale-Nausea+Vomiting: Stable | 64
  Scale-Nausea+Vomiting: Worsened | 2
  Symptom Scale-Pain: Improved | 62
  Symptom Scale-Pain: Stable | 29
  Symptom Scale-Pain: Worsened | 4
  Symptom - Dyspnoea: Improved | 12
  Symptom - Dyspnoea: Stable | 74
  Symptom - Dyspnoea: Worsened | 9
  Symptom - Insomnia: Improved | 53
  Symptom - Insomnia: Stable | 35
  Symptom - Insomnia: Worsened | 7
  Symptom - Appetite loss: Improved | 48
  Symptom - Appetite loss: Stable | 39
  Symptom - Appetite loss: Worsened | 8
  Symptom - Constipation: Improved | 46
  Symptom - Constipation: Stable | 45
  Symptom - Constipation: Worsened | 4
  Symptom - Diarrhoea: Improved | 18
  Symptom - Diarrhoea: Stable | 69
  Symptom - Diarrhoea: Worsened | 8
  Symptom - Financial difficulties: Improved | 17
  Symptom - Financial difficulties: stable: | 74
  Symptom - Financial difficulties: Worsened | 4

8. Secondary Outcome: Participant Counts in Response Categories Using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire For Pancreatic Cancer (EORTC-QLQ PAN26): Six Summary Scales
Description: The EORTC pancreatic cancer module is a validated tool intended for patients at all disease stages undergoing surgical resection, palliative surgical intervention, endoscopic palliation or palliative chemotherapy. The module includes 26 questions, organized into 7 scales and 10 individual item scores. All reported measures are transformed to a 0 to 100 scale. Six summary scales reported are: - Pancreatic Pain - Digestive Symptoms - Altered Bowel Habits - Hepatic Scale - Body Image - Sexuality Scores of 0 = optimal health state and 100 = worst possible health state. The best score on treatment is the best score from all post-baseline visits and is compared to the baseline. Responder categories: - Improved: >=MID decrease from baseline - Stable: no increase or decrease >MID - Worsened: >=MID increase from baseline MID = half the baseline standard deviation
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Groups:
- Nab-Paclitaxel Plus Gemcitabine: nab-Paclitaxel 125 mg/m^2 intravenous (IV) infusion administered over approximately 30-45 minutes on Days 1, 8, and 15, followed by gemcitabine 1000 mg/m^2 IV infusion over approximately 30 minutes on Days 1, 8, and 15 of each 28-day cycle. For participants who completed 6 cycles of nab-paclitaxel and gemcitabine the Investigator then determined the best option for the participant in the Investigator's Choice Period. - Continuation of nab-paclitaxel and gemcitabine therapy to disease progression or unacceptable toxicity OR - Chemoradiation therapy consisting of the concurrent use of capecitabine or gemcitabine with radiation according to institutional practice OR - Surgical intervention
Arm/Group | Nab-Paclitaxel Plus Gemcitabine
Number analyzed (Participants) | 95
Participants
  Pancreatic Pain Scale: Improved | 62
  Pancreatic Pain Scale: Stable | 33
  Pancreatic Pain Scale: Worsened | 0
  Digestive Symptom Scale: Improved | 49
  Digestive Symptom Scale: Stable | 36
  Digestive Symptom Scale: Worsened | 10
  Altered Bowel Habits Scale: Improved | 28
  Altered Bowel Habits Scale: Stable | 53
  Altered Bowel Habits Scale: Worsened | 14
  Hepatic Scale: Improved | 25
  Hepatic Scale: Stable | 66
  Hepatic Scale: Worsened | 4
  Body Image Scale: Improved | 22
  Body Image Scale: Stable | 50
  Body Image Scale: Worsened | 23
  Sexuality Scale: Improved | 31
  Sexuality Scale: Stable | 51
  Sexuality Scale: Worsened | 13

9. Secondary Outcome: Participant Counts in Response Categories Using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire For Pancreatic Cancer (EORTC-QLQ PAN26): Satisfaction With Health Care Scale
Description: The EORTC pancreatic cancer module is a validated tool intended for patients at all disease stages undergoing surgical resection, palliative surgical intervention, endoscopic palliation or palliative chemotherapy. The module includes 26 questions, organized into 7 scales and 10 individual item scores. The summary scale for Satisfaction with Health Care is reported. All reported measures are transformed to a 0 to 100 scale. Scores of 0 = not satisfied, worst possible health state and 100 = extremely satisfied, best possible health state. The best score on treatment is the best score from all post-baseline visits and is compared to the baseline to get the following responder categories. Responder categories: - Improved: >=MID increase from baseline - Stable: no increase or decrease >MID - Worsened: >=MID decrease from baseline MID = half the baseline standard deviation
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-Paclitaxel Plus Gemcitabine
Number analyzed (Participants) | 95
Participants
  Satisfaction with Health Care Scale: Improved | 42
  Satisfaction with Health Care Scale: Stable | 40
  Satisfaction with Health Care Scale: Worsened | 13

10. Secondary Outcome: Participant Counts in Response Categories Using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire For Pancreatic Cancer (EORTC-QLQ PAN26): 10 Individual Item Scores
Description: The EORTC pancreatic cancer module is a validated tool intended for patients at all disease stages undergoing surgical resection, palliative surgical intervention, endoscopic palliation or palliative chemotherapy. The module includes 26 questions, organized into 7 scales and 10 individual item scores. The 10 individual item scores are reported. All reported measures are transformed to a 0 to 100 scale. Scores of 0 = best possible health state and 100 = worst possible health state. The best score on treatment is the best score from all post-baseline visits and is compared to the baseline to get the following responder categories. Responder categories: - Improved: >=MID decrease from baseline - Stable: no increase or decrease >MID - Worsened: >=MID increase from baseline MID = half the baseline standard deviation
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Groups:
- Nab-Paclitaxel Plus Gemcitabine: nab-Paclitaxel 125 mg/m^2 intravenous (IV) infusion administered over approximately 30-45 minutes on Days 1, 8, and 15, followed by gemcitabine 1000 mg/m^2 IV infusion over approximately 30 minutes on Days 1, 8, and 15 of each 28-day cycle. For participants who completed 6 cycles of nab-paclitaxel and gemcitabine without disease progression or unacceptable toxicities, the Investigator then determined the best option for the participant in the Investigator's Choice Period.
Arm/Group | Nab-Paclitaxel Plus Gemcitabine
Number analyzed (Participants) | 95
Participants
  Abdominal Bloating: Improved | 50
  Abdominal Bloating: Stable | 42
  Abdominal Bloating: Worsened | 3
  Taste Changes: Improved | 20
  Taste Changes: Stable | 54
  Taste Changes: Worsened | 21
  Indigestion: Improved | 41
  Indigestion: Stable | 47
  Indigestion: Worsened | 7
  Flatulence: Improved | 47
  Flatulence: Stable | 37
  Flatulence: Worsened | 11
  Weight Loss: Improved | 36
  Weight Loss: Stable | 56
  Weight Loss: Worsened | 3
  Limb Weakness: Improved | 22
  Limb Weakness: Stable | 55
  Limb Weakness: Worsened | 18
  Dry Mouth: Improved | 37
  Dry Mouth: Stable | 45
  Dry Mouth: Worsened | 13
  Treatment Side-Effects: Improved | 8
  Treatment Side-Effects: Stable | 48
  Treatment Side-Effects: Worsened | 39
  Worry About Future Health: Improved | 42
  Worry About Future Health: Stable | 45
  Worry About Future Health: Worsened | 8
  Limits on Activity Planning: Improved | 42
  Limits on Activity Planning: Stable | 42
  Limits on Activity Planning: Worsened | 11

11. Secondary Outcome: Participants With Treatment Emergent Adverse Events (TEAEs)
Description: TEAEs are defined as any adverse event (AE) that begin or worsen on or after the start of study drug or procedure of the study period through the maximum duration of the period plus 28 days. The severity of AEs was graded based on National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0 and the scale: Grade 1 = Mild Grade 2 = Moderate Grade 3 = Severe Grade 4 = Life threatening Grade 5 = Death. Relation to study drug was determined by the investigator. A treatment-related TEAE is defined as TEAE which was considered to be related to one or both of the study drugs and reported as 'Suspected' on the case report form. AEs with a missing relationship were treated as 'treatment-related' in data summaries. IP (investigational product) refers to nab-Paclitaxel and/or Gemcitabine. "Related" TEAE refers to relation to study drug (IP).
Time Frame: Day 1 of study drug up to end of the study; up to 31.3 months
Population: The Treated population consists of all participants who received at least 1 dose of nab-paclitaxel or gemcitabine.
Measure: Count of Participants; unit: Participants
Groups:
- Nab-Paclitaxel Plus Gemcitabine (Induction Period): nab-Paclitaxel 125 mg/m^2 intravenous (IV) infusion administered over approximately 30-45 minutes on Days 1, 8, and 15, followed by gemcitabine 1000 mg/m^2 IV infusion over approximately 30 minutes on Days 1, 8, and 15 of each 28-day cycle.
  Six treatment cycles were planned.
- Nab-Paclitaxel Plus Gemcitabine (Overall): nab-Paclitaxel 125 mg/m^2 intravenous (IV) infusion administered over approximately 30-45 minutes on Days 1, 8, and 15, followed by gemcitabine 1000 mg/m^2 IV infusion over approximately 30 minutes on Days 1, 8, and 15 of each 28-day cycle.
  Overall includes nab-Paclitaxel plus Gemcitabine treatment cycles during the Induction Period, as well as the subset of participants who continued the regimen during the Investigator Choice Period.
Arm/Group | Nab-Paclitaxel Plus Gemcitabine (Induction Period) | Nab-Paclitaxel Plus Gemcitabine (Overall)
Number analyzed (Participants) | 106 | 106
Participants
  >= 1 TEAE | 105 | 105
  >=1 related TEAE | 102 | 103
  >=1 TEAE of severity grade 3 or higher | 85 | 90
  >=1 related TEAE of severity grade 3 or higher | 72 | 75
  >=1 serious TEAE | 38 | 39
  >= 1 related serious TEAE | 14 | 14
  >=1 TEAE leading to discontinuation of IP | 25 | 28
  >=1 related TEAE leading to discontinuation of IP | 15 | 18
  >=1 TEAE leading to dose reduction of IP | 69 | 72
  >=1 related TEAE leading to dose reduction of IP | 68 | 71
  >=1 TEAE leading to interruption of IP | 66 | 68
  >=1 related TEAE leading to interruption of IP | 48 | 50
  >= TEAE leading to death | 2 | 2
  >=1 related TEAE leading to death | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 of study drug up to end of the study; up to 31.3 months
Description: One participant was enrolled but not treated. The safety population consisted of participants who received at least one dose of nab-paclitaxel.
Groups:
- Nab-Paclitaxel Plus Gemcitabine (Induction Period): nab-Paclitaxel 125 mg/m^2 intravenous (IV) infusion administered over approximately 30-45 minutes on Days 1, 8, and 15, followed by gemcitabine 1000 mg/m^2 IV infusion over approximately 30 minutes on Days 1, 8, and 15 of each 28-day cycle.
Arm/Group | Nab-Paclitaxel Plus Gemcitabine (Induction Period) | Nab-Paclitaxel Plus Gemcitabine (Overall)
All-Cause Mortality (participants affected / at risk) | 42/106 | 67/106
Serious Adverse Events (participants affected / at risk) | 38/106 | 39/106
Other Adverse Events (participants affected / at risk) | 104/106 | 104/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nab-Paclitaxel Plus Gemcitabine (Induction Period) (N=106) | Nab-Paclitaxel Plus Gemcitabine (Overall) (N=106)
Blood bilirubin increased (Investigations) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Presyncope (Nervous system disorders) | 1 | 1
Obstructive uropathy (Renal and urinary disorders) | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 1
Jugular vein thrombosis (Vascular disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 2
Cardiac arrest (Cardiac disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Obstruction gastric (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 1 | 1
Generalised oedema (General disorders) | 1 | 1
Influenza like illness (General disorders) | 1 | 1
Malaise (General disorders) | 1 | 1
Pyrexia (General disorders) | 5 | 5
Cholangitis (Hepatobiliary disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 1
Cellulitis (Infections and infestations) | 2 | 2
Clostridium difficile colitis (Infections and infestations) | 1 | 1
Escherichia sepsis (Infections and infestations) | 1 | 1
Gastroenteritis Escherichia coli (Infections and infestations) | 1 | 1
Liver abscess (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 1
Neutropenic sepsis (Infections and infestations) | 2 | 2
Pancreas infection (Infections and infestations) | 1 | 1
Parainfluenzae virus infection (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 5 | 5
Sepsis (Infections and infestations) | 2 | 2
Peripancreatic fluid collection (Injury, poisoning and procedural complications) | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nab-Paclitaxel Plus Gemcitabine (Induction Period) (N=106) | Nab-Paclitaxel Plus Gemcitabine (Overall) (N=106)
Anaemia (Blood and lymphatic system disorders) | 49 | 49
Leukopenia (Blood and lymphatic system disorders) | 7 | 7
Lymphopenia (Blood and lymphatic system disorders) | 6 | 6
Neutropenia (Blood and lymphatic system disorders) | 44 | 45
Thrombocytopenia (Blood and lymphatic system disorders) | 25 | 27
Abdominal pain (Gastrointestinal disorders) | 19 | 19
Abdominal pain upper (Gastrointestinal disorders) | 9 | 10
Constipation (Gastrointestinal disorders) | 30 | 32
Diarrhoea (Gastrointestinal disorders) | 48 | 48
Dry mouth (Gastrointestinal disorders) | 7 | 7
Dyspepsia (Gastrointestinal disorders) | 7 | 8
Nausea (Gastrointestinal disorders) | 46 | 47
Stomatitis (Gastrointestinal disorders) | 20 | 20
Vomiting (Gastrointestinal disorders) | 30 | 30
Asthenia (General disorders) | 36 | 36
Chills (General disorders) | 18 | 18
Fatigue (General disorders) | 53 | 53
Influenza like illness (General disorders) | 7 | 8
Oedema peripheral (General disorders) | 45 | 47
Pain (General disorders) | 5 | 6
Pyrexia (General disorders) | 39 | 40
Upper respiratory tract infection (Infections and infestations) | 6 | 7
Alanine aminotransferase increased (Investigations) | 21 | 23
Aspartate aminotransferase increased (Investigations) | 16 | 17
Blood alkaline phosphatase increased (Investigations) | 14 | 16
Gamma-glutamyltransferase increased (Investigations) | 6 | 6
Neutrophil count decreased (Investigations) | 22 | 23
Platelet count decreased (Investigations) | 25 | 27
Weight decreased (Investigations) | 12 | 12
White blood cell count decreased (Investigations) | 14 | 14
Decreased appetite (Metabolism and nutrition disorders) | 46 | 46
Dehydration (Metabolism and nutrition disorders) | 11 | 11
Hyperglycaemia (Metabolism and nutrition disorders) | 12 | 12
Hyperkalaemia (Metabolism and nutrition disorders) | 6 | 6
Hypoalbuminaemia (Metabolism and nutrition disorders) | 11 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 14 | 14
Hypomagnesaemia (Metabolism and nutrition disorders) | 7 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 10 | 10
Iron deficiency (Metabolism and nutrition disorders) | 7 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 17
Bone pain (Musculoskeletal and connective tissue disorders) | 6 | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 12
Dizziness (Nervous system disorders) | 10 | 12
Dysgeusia (Nervous system disorders) | 32 | 33
Headache (Nervous system disorders) | 17 | 17
Neuropathy peripheral (Nervous system disorders) | 23 | 25
Paraesthesia (Nervous system disorders) | 11 | 11
Peripheral sensory neuropathy (Nervous system disorders) | 29 | 30
Anxiety (Psychiatric disorders) | 15 | 15
Depression (Psychiatric disorders) | 6 | 6
Insomnia (Psychiatric disorders) | 11 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 25
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 57 | 57
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 9 | 9
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 12
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 | 9
Hypotension (Vascular disorders) | 8 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is > 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 additional days. Investigator must delete confidential information before submission and defer publication to permit patent applications.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/43/NCT02301143/SAP_000.pdf
  • Study Protocol (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/43/NCT02301143/Prot_001.pdf